CLINICAL TRIAL: NCT02660424
Title: A Phase 2a Randomized, Double-blind, Placebo-Controlled, Crossover Study of the Efficacy and Safety of VX-150 in Subjects With Osteoarthritis of the Knee
Brief Title: A Study of the Efficacy and Safety of VX-150 in Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VX15-150-101
Record Dates: First submitted 2015-12-18; First posted 2016-01-21 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- VX-150, placebo (Experimental): Sequence 1: VX-150 in Treatment Period 1→washout→ placebo in Treatment Period 2
  Interventions: Drug: VX-150; Drug: Placebo
- placebo, VX-150 (Experimental): Sequence 2: placebo in Treatment Period 1→washout→ VX-150 in Treatment Period 2
  Interventions: Drug: VX-150; Drug: Placebo

INTERVENTIONS:
Drug: VX-150
Drug: Placebo

SUMMARY:
The Primary objective of this study is to evaluate the efficacy of VX-150 in the treatment of osteoarthritis pain

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.
* Subjects (male and female [of non-childbearing potential]) will be between the ages of 40 and 80 years, inclusive. Female subjects must have a negative pregnancy test at Screening and on Day 1 of each Treatment Period and must not be nursing; male subjects must not have a female partner who is pregnant or nursing.
* Body mass index (BMI) of 18.0 to 38.0 kg/m2, inclusive, and a total body weight of 50 to 150 kg.
* Ambulatory with osteoarthritis of the knee with symptoms for at least 6 months and pain on the majority of days for the past 30 days. Symptoms must include knee joint pain. In subjects with bilateral knee osteoarthritis, the more symptomatic knee will be considered the index knee.
* Radiographic evidence of at least one tibiofemoral osteophyte in the index knee within 12 months before the Day 1 Visit.
* WOMAC pain subscale score

Exclusion Criteria:

* History in the past 10 years of reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis, amyloidosis or fibromyalgia.
* History in the past 10 years of malignancy with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin or resected cervical atypia or carcinoma in situ.
* History of cardiac dysrhythmias requiring anti-arrythmia treatment(s).
* History of abnormal laboratory results ≥2.5 × upper limit of normal (ULN) indicative of any significant medical disease which in the opinion of the investigator would preclude the subjects participation in the study.
* A known or clinically suspected infection with human immunodeficiency virus or hepatitis B or C viruses.
* Other serious, acute or chronic medical or psychiatric illness that in the judgment of the investigator could compromise subject safety, limit the subject's ability to complete the study and/or compromise the objectives of the study.
* Either participated within 3 months in another investigational study in which the subject was exposed to study drugs or vaccines,or will participate concurrently in such study.
* History of drug or alcohol dependence in the past 3 years, or a positive test for drugs of abuse at the Screening Visit.
* Requires opioids for pain relief.
* Changed analgesic treatment regimen within 30 days of the Screening Visit.
* Received or plan to receive short acting hyaluronic acid, corticosteroid, or other intra-articular injections as follows:

  1. in the index knee within 3 months of the Screening Visit, or at any time during the study
  2. in any other joint within 4 weeks of the Screening Visit, or at any time during the study
* Received or plan to receive long acting hyaluronic acid or other intra-articular injections as follows:

  1. in the index knee within 6 months of the Screening Visit, or at any time during the study
  2. in any other joint within 4 weeks of the Screening Visit, or at any time during the study
* History of arthroscopic or open surgery within 12 months before the Screening Visit, or have a planned surgery during, or immediately after, study follow-up.
* History of joint replacement surgery in the index knee.
* Significant hip pain, ipsilateral to the index knee that may interfere with assessments of index knee pain.
* Clinical signs and symptoms of an active knee infection.
* Current use of a handicap assistance device (unilateral assistance device such as a cane is permitted).
* Started a new physical therapy, weight loss, or exercise program within 3 months of the Screening Visit, or are not willing to maintain a stable program during the course of the study.
* Lab abnormalities at the screening visit.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Western Ontario and McMaster Universities (WOMAC) osteoarthritis index pain subscale score at Day 14 | from baseline at Day 14

SECONDARY OUTCOMES:
Proportion of subjects with ≥50% reduction in WOMAC pain subscale at Day 14 | at Day 14
Change from baseline in total WOMAC score at Day 14 | at Day 14
Use of rescue medications [to be obtained by electronic diary and questionnaire] | Treatment periods1 (14 days) and 2 (14 days)
Safety and tolerability based on the incidence and type of adverse events (AEs),changes from baseline in clinically significant laboratory test results, and assessment of 12 lead electrocardiograms (ECGs) and vital signs at designated visits. | up to 12 weeks (duration of study)
Plasma PK parameters of prodrug, VX-150 and its primary metabolite: Cmax [maximum plasma concentrations] | Days 1,14 of each treatment periods
Plasma PK parameters of prodrug, VX-150 and its primary metabolite: Tmax [time to maximum plasma concentration] | Days 1,14 of each treatment periods
Plasma PK parameters of prodrug, VX-150 and its primary metabolite: AUC [area under the plasma concentration-time curve] | Days 1,14,16,18 of each treatment periods

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - San Diego, California
  - West Palm Beach, Florida
  - Marietta, Georgia
  - Valparaiso, Indiana
  - Wichita, Kansas
  - Bay City, Michigan
  - Las Vegas, Nevada
  - Hartsdale, New York
  - Duncansville, Pennsylvania
  - Providence, Rhode Island
  - Chattanooga, Tennessee
  - Danville, Virginia